CLINICAL TRIAL: NCT01547975
Title: Retrospective Analysis of Surgical Outcomes After Corneal Transplantation
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Hospital, Wei-Li Chen, MD, PhD, Assistant Professor, National Taiwan University Hospital, department of Ophthalmology., National Taiwan University Hospital
Other Study IDs: 201004004R
Record Dates: First submitted 2012-03-04; First posted 2012-03-08 (Estimated); Last update posted 2012-04-03 (Estimated); Status verified 2012-03

CONDITIONS: Corneal Transplantation
Keywords: surgical outcomes after corneal transplantation; Retrospective analysis; corneal transplantation

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Currently, no demographic and surgical results comparing different donor cornea sources were available in Taiwan. National Taiwan University Hospital (NTUH), as one of the largest tertiary medical centers in northern Taiwan, is now in charge of a big part of intense care for patients receiving corneal transplantation. With detailed medical record done of these patients during care in the ward and out-patient clinic, the investigators are competence for this meaningful program.

DETAILED DESCRIPTION:
An insufficient donor supply is a worldwide problem in organ transplantation. Even with corneal transplantations, the most widely performed transplantation, shortages and imbalances in donor supply is a global concern. In National Taiwan University Hospital (NTUH), the investigators performed over one hundred of corneal transplantations every year and the majority of donor corneas were from the eye bank in United States. Previous literature showed satisfactory results in corneal transplantation using foreign donor corneas compared with domestic corneas. However longer preservation time had associated with a statistically significant increased risk of persistence of the postoperative epithelial defect. On the other hand, longer storage times may allow better outcomes in high-risk grafts because of the depletion of donor T cells from the donor cornea into the storage media.

Currently, no demographic and surgical results comparing different donor cornea sources were available in Taiwan. NTUH, as one of the largest tertiary medical centers in northern Taiwan, is now in charge of a big part of intense care for patients receiving corneal transplantation. With detailed medical record done of these patients during care in the ward and out-patient clinic, the investigators are competence for this meaningful program.

ELIGIBILITY:
Inclusion Criteria:

* The patients who received corneal transplantation within full chart records

Exclusion Criteria:

* The patients have cognitive Impairment.
* No detail or unclear ophthalmologic record.
* Patients or their legal representative have no willing to accept this tracing study.

Max Age: 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The patients who received corneal transplantation within full chart records.
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2010-04; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Li Chen, MD,PhD, Study Chair — NTUH
Locations (1):
- National Taiwan University Hospital, department of Ophthalmology, Taipei, Taiwan, Taiwan